CLINICAL TRIAL: NCT04841265
Title: The Effect of Vitamin D Supplementation in Overweight and Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Loy See Ling, Senior Research Fellow, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIRB 2021/2055
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
Keywords: Vitamin D supplementation; Lipid profile; Vitamin D status; Birth outcomes; Pregnancy complications
MeSH Terms: conditions — Overweight; Obesity; Pregnancy Complications | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (Active Comparator): The Vitamin D3 (intervention) arm will receive a total of 800 IU vitamin D3 supplementation per day.
  Interventions: Dietary Supplement: Vitamin D3
- Control (No Intervention): The control arm will receive 400 IU vitamin D3 per day from routine antenatal multivitamin supplementation.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — The intervention arm will receive 400 IU vitamin D3 from routine antenatal multivitamin supplement tablet + 400 IU vitamin D3 daily until delivery.
  Arms: Vitamin D3

SUMMARY:
To understand the role of vitamin D supplementation on pregnancy outcomes and metabolic status in overweight and obese pregnant women.

DETAILED DESCRIPTION:
The effects of vitamin D supplementation on pregnancy outcomes and metabolic status of overweight and obese pregnant women remain uncertain. In particular, the dosage of vitamin D supplementation has not been defined in this high risk group of women. This study aims to examine whether oral supplement of vitamin D3 (cholecalciferol) in total dosage of 800 IU(prenatal multivitamin containing 400 IU vitamin D3 + 400 IU vitamin D3 alone) given to overweight and obese pregnant women since early pregnancy until delivery can improve maternal and neonatal outcomes, compared with those given prenatal multivitamin containing 400 IU vitamin D3 supplementation, a commonly given antenatal supplement in Singapore. The investigators' hypothesis is that higher dose vitamin D supplementation would lead to better outcomes in overweight and obese pregnant women. The investigators will conduct a two-arm, parallel non-blinded randomized controlled trial. Women with body mass index ≥25kg/m2 will be randomly assigned into groups with a 1:1 randomization ratio, receiving either 800 or 400 IU vitamin D3 supplementation. The study will be conducted at the antenatal clinics, KK Women's and Children's Hospital, Singapore. Measurements of serum 25-hydroxyvitamin D (25OHD), lipid profile and lifestyles information will be taken for all women at baseline (≤16 weeks gestation) and after three months of intervention (26-30 weeks gestation). All women will continue with the vitamin D3 supplementation until delivery. Primary outcomes include levels of maternal serum 25OHDconcentration and lipid profile at 26-30 gestation weeks as compared with the controls, adjusting for baseline measurements. Secondary outcomes include preeclampsia, gestational hypertension, gestational diabetes, glycaemic levels, caesarean section, gestational weight gain, preterm birth, low birth weight and small-for-gestational-age. This study will fill up the gap of knowledge regarding the role of vitamin D supplementation on pregnancy outcomes and metabolic status in overweight and obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation ≤16weeks (16 weeks + 6 days) upon intervention
2. Pre-pregnancy BMI ≥25 kg/m2
3. Aged 21-45 years
4. Willing and able to provide written, informed consent

Exclusion Criteria:

1. Having current or past hypo/hyperparathyroidism, hypercalciuria, hypercalcemia or osteomalacia
2. History of renal disease (including kidney stones and etc.), liver dysfunction, tuberculosis or sarcoidosis
3. Pre-existing diabetes mellitus or chronic hypertension
4. Taking lipid-lowering medicine
5. Gestational diabetes (as confirmed by oral glucose tolerance test) or gestational hypertensive disorder
6. Multiple pregnancy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Overweight and obese pregnant women
Enrollment: 274 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in maternal serum 25OHD concentration | Baseline, 26-30 gestational weeks
Change in maternal total cholesterol level | Baseline, 26-30 gestational weeks
Change in maternal HDL-cholesterol level | Baseline, 26-30 gestational weeks
Change in maternal LDL-cholesterol level | Baseline, 26-30 gestational weeks
Change in maternal triglyceride level | Baseline, 26-30 gestational weeks

SECONDARY OUTCOMES:
Incidence of preeclampsia | up to delivery
Incidence of gestational hypertension | Through pregnancy until delivery
Incidence of gestational diabetes | Through pregnancy until delivery
Fasting glucose level | 24-28 gestational weeks
1-hour post-load glucose level | 24-28 gestational weeks
2-hour post-load glucose level | 24-28 gestational weeks
Incidence of caesarean section | At delivery
Incidence of preterm birth (<37 weeks) | At delivery
Incidence of low birth weight (<2500g) | At delivery
Neonatal birth weight (g) | At delivery
Neonatal birth length (cm) | At delivery
Neonatal head circumference (cm) | At delivery
Incidence of admission to special care (including intensive care) during neonatal period | Within 28 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dr Loy See Ling, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No